CLINICAL TRIAL: NCT04012658
Title: A Registered Cohort Study on Wilson's Disease
Status: Recruiting | Type: Observational
Sponsor: Wan-Jin Chen (Other)
Responsible Party: Sponsor-Investigator, Wan-Jin Chen, The Vice-Director for the Department of Neurology, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH OF FMU[2019]197
Record Dates: First submitted 2019-07-06; First posted 2019-07-09 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Wilson's Disease
Keywords: Wilson's Disease; Nature history; Genetics
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with the genetic diagnosis of Wilson's Disease
  Interventions: Other: No intervention
- Asymptomatic Wilson's Disease carriers
  Interventions: Other: No intervention
- Relatives of Wilson's Disease patients or carriers
  Interventions: Other: No intervention
- Unrelated healthy controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of Wilson's Disease in a prospective multicenter natural history study, to assess the clinical, genetic, epigenetic features and biomarkers of patients with Wilson's Disease to optimize clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the genetic diagnosis of Wilson's Disease
* Asymptomatic Wilson's Disease carriers
* Relatives of Wilson's Disease patients or carriers
* Unrelated healthy controls
* Participants or Parent(s)/legal guardian(s) willing and able to complete the informed consent process

Exclusion Criteria:

* Participants are unable to comply with study procedures and visit schedule

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Wilson's Disease are diagnosed by the clinical and/or genetic features
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2039-12 (Estimated); Study Completion 2049-12 (Estimated)

PRIMARY OUTCOMES:
The change of Unified Wilson's Disease Rating Scale (UWDRS) | Up to 30years
  Disease severity will be assessed by application of the Unified Wilson's Disease Rating Scale (UWDRS), a clinical rating scale consists of three subscales. Higher UWDRS total scores indicate more severe disease.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, China